CLINICAL TRIAL: NCT00989937
Title: Double-Blind, Randomized, Placebo-Controlled, Cross-Over Pilot Study of Intranasal Oxytocin in Patients With Anxiety Disorder
Brief Title: Oxytocin Add-on Study for Stable Anxiety Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Break in funding
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David Feifel, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Oxytocin Anxiety
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Anxiety Disorders
Keywords: oxytocin
MeSH Terms: conditions — Anxiety Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): 20 IU BID for the first week, 40 IU BID for the following two weeks, one week washout, 3 week placebo trial
  Interventions: Drug: Oxytocin; Drug: Placebo
- Group 2 (Placebo Comparator): Three week placebo trial, one week washout, 20 IU BID for the fifth week, 40 IU BID for the following two weeks
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 20 IU BID or 40 IU BID
Drug: Placebo — 20 IU BID or 40 IU BID

SUMMARY:
The objective of the study is to compare the efficacy of intranasal oxytocin versus intranasal placebo to improve anxiety symptoms in patients with a variety of anxiety disorders.

DETAILED DESCRIPTION:
Anxious patients treated with even the best currently available anti-anxiety drugs continue to experience significant symptoms.

A variety of basic science, animal studies, and human studies support the idea that the neuropeptide oxytocin may be effective against anxiety in humans. For example, plasma oxytocin levels may function as an index of central serotonin (5-HT) function in human subjects, and serotonin is well-known to be involved in clinical anxiety disorders. Since oxytocin is released directly from limbic-hypothalamic cells, this response presumably represents a direct central assessment of 5-HT response in limbic-hypothalamus (Lee 2003). In animal models, Ring 2006 examined the effects of oxytocin on both behavioral and autonomic parameters of the anxiety response in male mice using three pharmacologically validated preclinical models of anxiety: the four-plate test (FPT), elevated zero maze (EZM), and stress-induced hyperthermia (SIH). The results from this study provide specific behavioral and autonomic evidence of anxiolytic-like effects for oxytocin. In primates, Emiliano et al 2007 found support for the idea that that SSRIs' therapeutic effects on social affiliation and anxiety may be mediated in part through components of the oxytocin system. Human studies include Kosfeld et al (2005), who demonstrated that oxytocin administered intranasally to healthy human subjects in a double-blind, placebo controlled study increased levels of trust. As well, Kirsch et al (2005) showed that intranasal oxytocin reduced activation of brain circuits involved in fear in human subjects. Finally, Scantamburlo (2007) showed a significant negative correlation between oxytocin and the scored symptoms depression and anxiety. These studies clearly suggest the potential utility of OTR agonism as a therapeutically relevant mechanism of action for novel anxiolytics in both sexes.

Each subject will be enrolled for 6 week treatment period after a screening phase. Study procedures involve weekly clinic visits as an outpatient. Forty patients will be randomly assigned to either 40 International Units (IU) oxytocin twice daily or vehicle placebo. After 3 weeks, treatments will be crossed over such that subjects that received oxytocin will receive placebo and vice versa. The study ratio is 1:1. Dose of oxytocin is based upon previous studies in humans showing improvement in psychiatric populations related changes in behavior and brain function (Kosfeld et al, 2005; Kirsch 2005; Heinrich M 2003).

The total study duration for each individual subject will be approximately 7 weeks, which includes up to 21-day screening/wash-out period, a baseline (randomization) visit, three week treatment period, 1 week washout, baseline, and three weeks cross over treatment.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Generalized Anxiety Disorder (GAD), Social Anxiety Disorder (SAD), Post-traumatic stress disorder, or Anxiety Disorder NOS, confirmed by a semi-structured interview with the Structured Clinical Interview for DSM-IV Axis Disorders-Modified-Patient Edition (SCID).
2. HAM-A total score ≥15 with Item 1 (anxious mood) and Item 2 (tension) scores ≥2 at randomization.
3. Have a Clinical Global Impressions-Severity (CGI-S) scale score of at least 4 (moderately ill) at baseline;
4. Must be able to communicate effectively with the investigator and study coordinator and have the ability to provide informed consent.
5. Must demonstrate an acceptable degree of compliance with medication and procedures in the opinion of the investigator
6. Adult men or women, 18 years of age or older.
7. Laboratory results, including serum chemistries, hematology, and urinalysis, must show no clinically significant abnormalities (clinically significant is defined as laboratory values requiring acute medical intervention, indicating a serious medical illness, or requiring further medical evaluation in the judgment of the investigator). In addition, there must be no clinical information that, in the judgment of a physician, should preclude a subjects' participation at study entry.
8. Must be able to use nasal spray
9. Must be able to communicate effectively with the investigator and study coordinator.
10. Patients may be taking a variety of medications for anxiety at the time of enrollment, or may be receiving no medication treatment, but must be stable on their particular regiment for 3 weeks. If the subject is in the process of changing medications, enrollment will be deferred

Exclusion Criteria:

1. Are pregnant or are breastfeeding
2. A urine drug screen at screening that is positive for recent use of illegal drugs or alcohol
3. Any active medical condition that in the opinion of the investigator will interfere with the objectives of the study
4. For any reason the investigator considers the subject to be an unsuitable candidate to receive Oxytocin or believes the subject would be non-compliant with taking the study drug or study procedures.
5. Subjects with a score greater than 1 on question #3 "Suicide". suicidal is excluded.
6. Subjects with a total score greater than 17 on the 21 item scale, HAMD, are excluded from participating.
7. Subjects with a diagnosis of Obsessive Compulsive Disorder, a psychotic disorder, bipolar disorder, or with substance abuse or dependence in the prior 6 months will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Feifel, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Period: Overall Study
Arm/Group | All Participants
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Total Score on the Hamilton Anxiety Scale (HAM-A)
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Clinical Global Impression - Severity of Illness (CGI-S
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Social Phobia Inventory (SPIN)
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: The State-Trait Anxiety Inventory (STAI)
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: The Profile of Mood States (POMS)
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Sheehan Disability Scale (SDS)
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Arizona Sexual Experience Scale (ASEX)
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Hamilton-Depression Scale (HAM-D)
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Reading Trust in the Mind in the Eyes Test (RTET)
Time Frame: Visits 1, 4, 5, 8
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Childhood Trauma Questionnaire [CTQ]
Time Frame: Visit 1 (only once)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Global Assessment of Functioning (GAF)
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes